CLINICAL TRIAL: NCT04954508
Title: The Hug-up Test: A New, Sensitive Diagnostic Test for Supraspinatus Tears
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014156
Record Dates: First submitted 2021-07-05; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- P: patients suffering form shoulder pain and/or weakness or dislication
  Interventions: Diagnostic Test: The hug-up test; Diagnostic Test: EC test; Diagnostic Test: FC test; Diagnostic Test: Neer impingement sign; Diagnostic Test: Hawkins-Kennedy impingement sign; Diagnostic Test: diagnostic arthroscopy

INTERVENTIONS:
Diagnostic Test: The hug-up test — It is a new physical test used to detect supraspinatus tear
Diagnostic Test: EC test — It is a traditional physical test used to detect supraspinatus tear
Diagnostic Test: FC test — It is a traditional physical test used to detect supraspinatus tear
Diagnostic Test: Neer impingement sign — It is a traditional physical test used to detect supraspinatus tear
Diagnostic Test: Hawkins-Kennedy impingement sign — It is a traditional physical test used to detect supraspinatus tear
Diagnostic Test: diagnostic arthroscopy — The arthroscopic operation involved complete inspection of the supraspinatus. Supraspinatus tears were categorized as fullthickness tears (FTTs), which were classified as small (≤1 cm), moderate (≤3 cm), large (≤5 cm), and massive (>5 cm), on the basis of the largest dimension, and partial-thickness tears (PTTs), which were classified as bursal-sided, articular-sided,and intra-tendinous. Other combined diseases including acromioclavicular joint derangement, infraspinatus lesions, subscapularis lesions, superior labrum anterior and posterior (SLAP) lesions, biceps disorders, and Bankart lesions were recorded as well to assess the specificity of the tests.

SUMMARY:
We developed a new test, the "hug-up test," wherein elevation is resisted as the palm is held on the opposite shoulder with the elbow held in maximal anterior translation. The purpose of this study was to describe the hug-up test and compare it with other conventional tests used for diagnosing supraspinatus tears.

DETAILED DESCRIPTION:
The supraspinatus tendon is the most commonly affected tendon in rotator cuff tears. Early detection of a supraspinatus tear using an accurate physical examination is, therefore, important. However, the currently used physical tests for detecting supraspinatus tears are poor diagnostic indicators and involve a wide range of sensitivity and specificity values. Therefore, the aim of this study was to establish a new physical test for the diagnosis of supraspinatus tears and evaluate its accuracy in comparison with conventional tests.

Between November 2012 and January 2014, 200 consecutive patients undergoing shoulder arthroscopy were prospectively evaluated preoperatively. The hug-up test, empty can (EC) test, full can (FC) test, Neer impingement sign, and Hawkins-Kennedy impingement sign were used and compared statistically for their accuracy in terms of supraspinatus tears, with arthroscopic findings as the gold standard. Muscle strength was precisely quantified using an electronic digital tensiometer.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo an arthroscopic procedure for a diagnosis related to shoulder pain and/or weakness or dislocation by one of the senior authors from November 2012 to January 2014

Exclusion Criteria:

* Patients with a history of shoulder surgery, upper extremity fractures, and bilateral shoulder diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 200 consecutive patients scheduled to undergo an arthroscopic procedure for a diagnosis related to shoulder pain and/or weakness or dislocation by one of the senior authors.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
patients' self-reported pain | immediately after the test
  Pain experienced during the Neer impingement and Hawkins-Kennedy impingement tests and weakness during the EC test and the FC test were considered positive results.
diagnostic arthroscopy | during the arthrosocpic procedure
  The arthroscopic operation involved complete inspection of the supraspinatus. Supraspinatus tears were categorized as fullthickness tears (FTTs), which were classified as small (≤1 cm), moderate (≤3 cm), large (≤5 cm), and massive (>5 cm), on the basis of the largest dimension, and partial-thickness tears (PTTs), which were classified as bursal-sided, articular-sided,and intra-tendinous. Other combined diseases including acromioclavicular joint derangement, infraspinatus lesions, subscapularis lesions, superior labrum anterior and posterior (SLAP) lesions, biceps disorders, and Bankart lesions were recorded as well to assess the specificity of the tests.the supraspinatus. Supraspinatus tears were categorized as fullthickness tears (FTTs), which were classified as small (≤1 cm), moderate (≤3 cm), large (≤5 cm), and massive (>5 cm), on the basis of the largest dimension, and partial-thickness tears (PTTs), which were classified as bursal-sided, articular-sided,

CONTACTS AND LOCATIONS:
Overall Officials: Yulei Liu, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No